CLINICAL TRIAL: NCT06501924
Title: Clinical Study of DA-002 and DA-005 As a Treatment for Hair Loss
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Applied Biology, Inc. (Industry)
Collaborators: Follea International Limited (Industry); Daniel Alain, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DA-005
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Androgenetic Alopecia; Female Pattern Baldness; Male Pattern Baldness
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- DA-005 (Experimental): Oral Botanical Supplement HIF-1a inhibitor
  Interventions: Dietary Supplement: DA-005; Other: Placebo Topical Solution
- Topical Minoxidil 5% (Active Comparator): Topical Minoxidil 5%
  Interventions: Drug: Topical minoxidil 5%; Dietary Supplement: Placebo Oral Tablet
- DA-002 (Experimental): Topical Alpha 1 Agonist
  Interventions: Drug: DA-002; Dietary Supplement: Placebo Oral Tablet

INTERVENTIONS:
Dietary Supplement: DA-005 — Oral Botanical Supplement HIF-1a inhibitor
  Other Names: Daniel Alain Botanical Supplement Treatment for Hair Loss
  Arms: DA-005
Drug: Topical minoxidil 5% — Topical minoxidil 5%
  Arms: Topical Minoxidil 5%
Drug: DA-002 — Topical Alpha 1 Agonist (GRAS)
  Arms: DA-002
Dietary Supplement: Placebo Oral Tablet — Placebo Oral Tablet
  Arms: DA-002; Topical Minoxidil 5%
Other: Placebo Topical Solution — Placebo Topical Solution
  Arms: DA-005

SUMMARY:
The primary objective of the study is to assess the safety and efficacy of DA-005 and DA-002 as a treatment for hair loss (androgenetic alopecia).

DETAILED DESCRIPTION:
DA-005 is a botanical supplement with demonstrated HIF-1a inhibitory action. The ingredients were tested in-vitro and have demonstrated the HIF-1a inhibitory effect. The primary aim of the study is to compare DA-005 to topical minoxidil in the treatment of hair loss (also known as androgenetic alopecia).

DA-002 is a topical alpha 1 agonist. The ingredients were tested in-vitro and have demonstrated hair growth effects. The secondary aim of the study is to compare DA-002 to topical minoxidil in the treatment of hair loss (also known as androgenetic alopecia).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Diagnosed with androgenetic alopecia
* Willing and able to apply the treatment as directed, comply with study
* Otherwise healthy
* Able to give informed consent

Exclusion Criteria:

* A medical history that may interfere with study objectives
* Women who are pregnant, lactating, or planning to become pregnant during the study period
* Subjects who have experienced a clinically important medical event within 90 days of the visit (e.g., stroke, myocardial infarction, etc)
* Subjects who have known allergies to any excipient in DA-002 or DA-005
* Subjects who are currently participating in another clinical study or have completed another clinical study with an investigational drug or device in the treatment area within 30 days prior to study treatment initiation
* Subjects who have used any topical prescription medications in the treatment area within 30 days prior to study treatment initiation
* Subjects who have had a dermatological procedure such as surgery in the treatment area within 30 days prior to study treatment initiation
* Subject is unable to provide consent or make the allotted clinical visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-10-17 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Target Area Hair Counts | Week [0,12]
  Target Area Hair Counts
Target Area Hair Counts | Week [0,24]
  Target Area Hair Counts

CONTACTS AND LOCATIONS:
Overall Officials: Andy Goren, MD, Study Director — University of Rome G. Marconi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Daniel Alain, Inc. - Updated Study Information — http://www.danielalain.com